CLINICAL TRIAL: NCT04764344
Title: A Single Center, Randomized Controlled Prospective Double-blinded Trial Comparing Haloperidol to Standard Ondansetron Therapy for Control of Nausea and Vomiting in the Emergency Department
Brief Title: Haloperidol for the Treatment of Nausea and Vomiting in the ED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Western Michigan University School of Medicine (Other)
Responsible Party: Principal Investigator, Jessica J McCoy, MD FACEP, Clinical Associate Professor, Western Michigan University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WMed-2020-0690
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Vomiting; Nausea; Abdominal Pain; Cannabis Use
MeSH Terms: conditions — Vomiting; Nausea; Abdominal Pain | interventions — Haloperidol; Ondansetron

STUDY DESIGN:
Intervention Model Description: This is a single-center prospective randomized double-blinded non-inferiority trial with potential assessment of superiority comparing haloperidol to ondansetron for the treatment of nausea and vomiting.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Treatment allocations will be revealed only after study completion, unless there is concern for a serious adverse event in which case treatment team and patient will be unblinded. Interim analysis will be performed at 150 participants to evaluate for effectiveness and power
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Haloperidol (Experimental): 2.5 mg of IV haloperidol diluted to a final concentration of 5 mL with 0.9% sodium chloride
  Interventions: Drug: Haloperidol
- Ondansetron (Active Comparator): 4 mg of IV ondansetron diluted to a final concentration of 5 mL with 0.9% sodium chloride
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Haloperidol — 2.5mg of IV haloperidol will be diluted to 5ml with 0.9% NS and given over 2 minutes IVP
  Other Names: Haldol
  Arms: Haloperidol
Drug: Ondansetron — Ondansetron
  Arms: Ondansetron

SUMMARY:
Single center, double-blind, randomized, controlled trial in patients who present to the emergency department (ED) with a chief complaint of nausea or vomiting. A total of 300 patients age 18-55 presenting to the emergency department with chief complaint of nausea or vomiting will be enrolled from February 2021 - February 2022. Patients will be randomized and symptom levels will be recorded at 30, 60, 90, minutes. Follow-up will be performed by telephone at 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* presenting to the emergency department with chief complaint of nausea or vomiting

Exclusion Criteria:

* abnormal blood pressure (>200/100mmHg or <90/40mmHg),
* fever (>100.4F),
* acute trauma,
* QT > 450ms on cardiac monitor,
* altered mental status (GCS < 15),
* chest pain,
* known allergy to haloperidol or ondansetron,
* Parkinson's disease,
* pregnancy or lactation,
* use of any antiemetic in the previous 8 hours,
* nausea and vomiting associated with vertigo,
* prisoners or any wards of the state.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | from enrollment to 30, 60, and 90 minutes after drug administration
  Mean change in visual analog scale (VAS) of self-rated nausea severity

SECONDARY OUTCOMES:
Analgesia | 0, 30, 60, 90 minutes
  Measurement of analgesia graded based on a self-reported validated 10 point visual analog scale (VAS)
Efficacy in marijuana users | Baseline (time 0)
  Marijuanna use will be documented and quantified
QT prolongation | Baseline (time 0) and 90 minutes
  QT will be measured on the cardiac monitor
Incidence of side-effects | 0, 30, 60, 90 minutes and 24 hours
  Inquiry about side effects

CONTACTS AND LOCATIONS:
Overall Officials: Jessica McCoy, MD, Principal Investigator — Western Michigan University School of Medicine
Locations (1):
- Bronson Methodist Hospital, Kalamazoo, Michigan, United States

DOCUMENTS (1):
  • Informed Consent Form (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/44/NCT04764344/ICF_000.pdf